CLINICAL TRIAL: NCT01357382
Title: The ACT-OUT Trial: ACTivity OUTcomes Based on the Consumption of a High Carbohydrate or High Fat Diet in Patients With Metabolic Syndrome
Brief Title: The ACT-OUT Trial: ACTivity OUTcomes Based on High Carbohydrate or High Fat Diet in Metabolic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Sammy Chan, Healthy Heart Program, St. Paul's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02652
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-04

CONDITIONS: Metabolic Syndrome
Keywords: low fat diet; low carbohydrate diet
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low fat diet (No Intervention): replace high fat, energy dense foods with foods rich in whole grains, fruits and vegetables. The macronutrient distribution of this diet will be approximately 55% carbohydrate, 15% protein and 30% fat. Individuals will also be instructed to reduce sodium intake to < 2300 mg / day and in individuals with hypertension, < 1500 mg / day.
- low carbohydrate diet (Experimental): restrict carbohydrate consumption to < 20 grams / day while not restricting caloric intake. Participants will be encouraged to consume vegetables with low carbohydrate content every day including 2 cups of salad greens and 1 cup of vegetables 'that grow above the ground' to increase their salt intake by consuming two cups of broth , ½ teaspoon of salt, or tablespoons of salt daily
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet — restrict carbohydrate consumption to < 20 grams / day while not restricting their caloric intake. Participants will be encouraged to consume vegetables with low carbohydrate content every day including 2 cups of salad greens and 1 cup of vegetables 'that grow above the ground' increase their salt intake by consuming two cups of broth , ½ teaspoon of salt, or tablespoons of salt daily
  Arms: low carbohydrate diet

SUMMARY:
Current obesity prevention emphasizes caloric restriction and avoidance of high fat foods. The result is an approach that replaces dietary fat with carbohydrates. There has, however, since been an obesity epidemic with an increased prevalence of metabolic syndrome (MetS) and type II diabetes. Negative results from trials of low fat diets for weight loss, prevention of heart disease and malignancies are consistent with the inadequacy of low fat/high carbohydrate approach. One of the findings of trials comparing low fat, calorie reduced diets to ad lib carbohydrate restricted diets is that subjects randomized to a low carbohydrate intake lose more weight despite equivalent intake. This equates to a 200 kcal/day greater weight loss on a carbohydrate restricted diet. Some investigators have speculated the metabolic advantage of carbohydrate restriction is due to increased energetic costs of gluconeogenesis. Alternatively, carbohydrate restriction is associated with increases in spontaneous physical activity.

This protocol has three aims. First, adherence to a carbohydrate restricted diet in subjects with metabolic syndrome will cause an increase in spontaneous physical activity, independent of weight changes. Second, cardiometabolic risk factors (ApoB, TG, HDL, blood pressure, CRP) will show greater improvement on a carbohydrate restricted diet compared to a low-fat, high carbohydrate diet. Finally the investigators will interview a sub-sample of participants to better understand quality of life issues with respect to the dietary assignment or lifestyle intervention.

The investigators will recruit 72 participants with MetS, from the Metabolic Syndrome Program at St. Paul's Hospital, Vancouver. Individuals will be randomized to either a low-carbohydrate diet or a calorie restricted, low fat diet and followed for 6 months. The investigators will measure body composition with bioelectrical impedance at baseline, 3 and 6 months. The investigators will also examine cardiometabolic changes due to the standard lifestyle intervention compared to the carbohydrate restricted treatment. The investigators will examine blood pressure, triglycerides, LDL-chol, HDL-chol, C-reactive protein, apolipoprotein B, glucose, insulin, hemoglobin A1c and leptin at baseline, 3 and 6 months. The investigators will use accelerometers to assess changes in physical activity. The investigators will use three-way repeated-measures ANOVA, with changes in body weight and insulin levels as covariates in the model with time as the repeated factor for statistical analyses.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE:

   Current obesity prevention emphasizes increasing physical activity and a low-fat, calorie restricted diet to produce a negative caloric balance. Caloric restriction is associated with decreases in energy expenditure. The other mainstay of obesity prevention increasing levels of physical activity is associated with greater caloric intake. Failure of the eat less-exercise more strategy is evident with epidemic of obesity, metabolic syndrome (MetS) and type II diabetes. Moreover, the displacement of dietary fat in the diet has led to compensatory increases in carbohydrate intake that is associated with untoward metabolic effects.

   Carbohydrate restricted diets are controversial despite benefits of this approach. The controversy stems from a compensatory increase in dietary fat intake associated with carbohydrate restriction and fears that greater fat intake increases risk of cardiovascular disease. Carbohydrate restriction decreases insulin resistance and ameliorates MetS. This protocol aims to establish a greater evidence base for carbohydrate restricted diets as a therapeutic option for MetS. The investigators will review current knowledge with respect to: (i) obesity and insulin resistance in Canada, (ii) positions of major medical organizations (iii) shortcomings of the current obesity prevention paradigm (iv) why carbohydrate restricted diets work.

   1.1) Obesity and insulin resistance in Canada In the 1980s low fat, caloric restricted diets became the cornerstone of dietary advice to reduce obesity. This approach successfully reduced the percent of calories from fat with a consequential increase in carbohydrate consumption. In the ensuing years, obesity become epidemic. In Canada, the prevalence of obesity (BMI ≥ 30 kg/m2) increased from 10% in 1970s to 23% in 2004 with an additional 36% considered overweight (BMI 25-29.9). As obesity is a risk factor for MetS and type II diabetes, the prevalence of these disorders has also reached epidemic proportions. Approximately 2 million Canadians were living with diabetes in 2007 and by 2012 it is estimated that 2.8 million Canadians will be living with diabetes. First Nations communities have been especially hard hit, with a prevalence 3-4 times higher and a younger age of onset than non-First Nations individuals. Novel chronic disease prevention strategies are needed to address this crisis.

   Insulin resistance underpins the pathophysiology of obesity, Insulin resistance is a condition in which normal amounts of insulin are inadequate to produce a normal insulin response from fat, muscle and liver cells. As a result, insulin resistant individuals have both elevated blood glucose, fasting insulin and secrete greater amounts of insulin in response to dietary carbohydrate. This compensatory hyperinsulinemia is associated with adverse effects in tissues which retain their sensitivity to insulin. Elevated blood glucose levels are associated with advanced glycation end products, reactive oxygen species and low grade inflammation. These exposures are associated with increased risk of cardiovascular disease & diabetes. Despite the evidence associating elevated insulin levels to atherogenic changes in the vasculature, it remains a matter of controversy as to whether persistently elevated insulin levels are pathogenic.

   The diagnosis of MetS represents an entry-point for disease prevention efforts in individuals with diabetes and cardiovascular disease. MetS is defined as a high waist circumference in addition to two of the following: high triglycerides, low HDL and elevated blood pressure. Other pathophysiologic changes are also observed including low grade inflammation, increased uric acid, prothrombotic state, elevated ApoB, small dense atherogenic LDL and endothelial dysfunction.

   First line treatment for MetS is weight loss leading to reductions in insulin resistance. Intensive lifestyle interventions reduce diabetes in high risk subjects. Most lifestyle interventions for MetS are predicated on the hypothesis that individuals can initiate and maintain weight loss by restricting calories and increasing physical activity. The Diabetes Prevention Program showed that intensive intervention including a low-fat calorie reduced diet and increase in physical activity was associated 1.5 kg/m2 decrease in BMI and a 58% reduction in incidence of diabetes in individuals at high risk of diabetes. Less intensive interventions are associated with more modest changes. A study of nutritional counselling was associated with a 0.4 kg/m2 decrease in BMI. Thus, lifestyle interventions which emphasize 'eating less or exercising more have limited value. The optimal diet for subjects with MetS has not been examined with hard end-points. Small trials have compared carbohydrate restricted diets and low fat diets using surrogate markers. A trial of severely obese subjects found greater weight loss and greater improvements in lipid levels and hemoglobin A1c on carbohydrate restricted diet than low fat/calorie restricted diets. In a study of adults with MetS, those randomized to the carbohydrate restriction had greater weight loss, lower triglycerides and lower insulin levels than individuals on a calorie restricted, low fat diet. These results are consistent with a meta-analysis where carbohydrate restricted diets were associated with improvements in atherogenic dyslipidemia, greater weight loss and better compliance than low fat, calorie restricted diets. These studies highlight the advantages of carbohydrate restriction.

   1.2) Fat, sugar and positions of major medical organizations One of the principal barriers to the widespread implementation of carbohydrate restricted diets is the fear that increase in saturated fat consumption with its association with increase in LDL-chol, will result in greater risk of cardiovascular disease (CVD). This diet-heart hypothesis has formed the cornerstone of dietary advice for prevention of chronic disease. The avoidance of saturated fat has led to general avoidance of dietary fat. There is weak and contradictory evidence that both saturated fat and dietary fat restriction are associated with health benefits. The largest test of the diet-heart hypothesis was the Women's Health Initiative (WHI). This study randomized women to either a low saturated fat diet or a regular diet. After 8 years, women randomized to the low fat diet had lower LDL-chol but no decrease in CVD mortality, incidence of breast or colorectal cancer. Consistent with the results of the WHI, a meta-analysis which included 347,747 subjects found no relationship between saturated fat intake and CVD.

   While most experts would agree that it's too early to vindicate saturated fat as the foremost dietary evil, evidence is accumulating highlighting the obesigenic and atherogenic nature of refined carbohydrates. A trial aiming to decrease sweetened beverage consumption found the intervention group had 7.7% less overweight and obese children than controls. In NHANES (2006), consumption of added sugar was associated with higher triglycerides and lower HDL. A prospective study of Dutch adults found that replacing 5% of calories from saturated fat with high glycemic carbohydrates was associated with a 33% increase in risk of myocardial infarction.

   The current state of scientific confusion over the health effects of (refined) carbohydrates is reflected in the diversity of dietary recommendations. American Diabetes Association (ADA) dietary guidelines have suggested that carbohydrate restricted diets are an option for weight loss for up to 1 year. In contrast, Canadian Diabetes Association recommends a diet with 45%-60% of calories from carbohydrate with a sucrose intake up to 10% of daily intake. The contradictory nature of these positions highlights the need for more research into the health effects of carbohydrate restricted diets. The endorsement of carbohydrate restriction by ADA suggests that these diets are valid therapeutic options.

   1.3) Shortcomings of the traditional obesity prevention paradigm The current obesity prevention paradigm emphasizes caloric reduction and/or increased physical activity to produce negative caloric balance. While physical activity has established benefits, increasing physical activity as a weight loss strategy has met with disappointing results. Observational studies associating high levels of physical activity with lower adiposity are difficult to interpret as individuals with higher physical activity also benefit from other (unmeasured) health promoting behaviours. In randomized trials, physical activity interventions have shown equivocal results with respect to weight loss. The physiologic limitation of this approach is that it is difficult to augment physical activity without a compensatory increase in dietary intake. In studies where physical activity is directly supervised and in the absence of a compensatory increase in caloric intake, physical activity has been associated with weight loss < 3% of initial body weight. In physical activity interventions of lower intensity, results are less promising. A meta-analysis of school based physical activity interventions in youth found no effect on BMI. The ineffectiveness of physical activity as a means of weight loss is reflected in the American Heart Association and American College of Sports of Sports Medicine position statements where they recommend 60-90 minutes of moderate intensity activity/day to lose or maintain weight loss. Not surprisingly, there is a very low prevalence of individuals who are moderately active for 60-90 minutes/day in the general population. Ironically, insulin resistant individuals who would reap the greatest health benefits from physical activity may have a reduced physiologic tolerance for it as insulin resistance has been associated with reduced exercise tolerance through reversible changes in muscle mitochondria, reduced VO2 max and possibly other mechanisms.

   The failure of low fat, calorie restricted diets to curb the prevalence of obesity is exemplified by the WHI. After 7.5 years of follow-up, the women randomized to the low fat group decreased their weight by 0.8 kg but had a 1 cm increase in waist circumference despite a reported decrease in caloric intake of 360 calories. Weight loss in the low fat group was not different than women in the control group, who were consuming a typical American diet. Calorie restricted diets emphasize the avoidance of energy dense foods high in dietary fat. While avoidance of dietary fat has intuitive appeal, calorie restriction is associated with a corresponding decrease in energy expenditure, in effect, stimulating a starvation response. The compensatory decrease in energy expenditure is associated with a plateauing of weight loss, an increased desire to eat and weight gain.

   Low fat/high carbohydrate diets require weight loss to produce positive metabolic effects. This dependence on weight loss for health benefits combined with the inevitable rebound weight gain associated with this dietary strategy has the potential to worsen metabolic markers over the long term. The untoward metabolic changes associated with a high carbohydrate intake are particularly deleterious in individuals with MetS. This contrasts with the physiologic effects of carbohydrate withdrawal in insulin resistant subjects that mirrors reversal of MetS. In addition to improvements of MetS, carbohydrate restricted diets are associated with less dense and therefore less atherogenic LDL particles and decreases in inflammatory markers.

   A final limitation of the current obesity prevention paradigm is that macronutrients (fat, protein and carbohydrates) are assumed to have equivalent metabolic effects. The investigators will review metabolic effects of macronutrients relating to the insulin response and energy balance. Carbohydrates are potent secretagogues of insulin that is the primary regulator of adipose tissue metabolism and partitions dietary energy into either storage (higher insulin) or oxidation (lower insulin). Mice genetically engineered to lack the insulin receptor on fat cells consume more calories per gram of body weight but are resistant to obesity. In type II diabetics, administrations of exogenous insulin or drugs which stimulate insulin release from the pancreas are associated with weight gain. Dietary fat has no effect on insulin secretion but delays gastric emptying. Dietary protein lowers the glucose response to insulin 2-3 times more effectively than dietary fat and plays an important role in appetite suppression and potentially weight regulation. The addition of dietary fat, protein and fiber to dampen the untoward effects of dietary carbohydrate in a meal is the concept behind the glycemic index. Low glycemic index diet may be of less relevance to type II diabetics, however, as the effect of dietary fat and protein in blunting glucose responses is attenuated or absent. If obesity prevention is indeed evidence base then there are only two tools left in the public health arsenal, bariatric surgery or carbohydrate restriction.

   1.4) Why do carbohydrate restricted diets work? There are at least two physiologic characteristics of carbohydrate restricted diets which contribute to weight loss. First, ad lib carbohydrate restricted diets have been associated with spontaneous reductions in caloric intake. Second, these diets are associated with greater weight loss per calorie than low-fat diets with an unexplained caloric deficit of about 200 kcal/day. The preferential weight loss of carbohydrate restricted diets was termed 'the metabolic advantage'. The concept of a metabolic advantage associated with carbohydrate restricted diets has been controversial among experts. While there is evidence supporting its existence in animal models and in humans, this phenomena remains poorly understood.

   Ad lib carbohydrate restricted diets are often associated with spontaneous decreases in caloric intake. This is caused by the insulin lowering effects of carbohydrate restricted diets as high insulin levels have been associated with partitioning of metabolic fuels into adipose tissue and greater food intake. A trial of obese subjects found that those consuming a carbohydrate restricted diet had nearly a 30% decrease in fasting insulin levels and a 570 kcal decrease in energy intake. Thus lower insulin levels are a key mediator between lower carbohydrate consumption and weight loss. A study in men found that 70% of the variability in weight loss from a carbohydrate restricted diet was explained by changes in fasting insulin.

   A number of trials have shown a metabolic advantage of carbohydrate restricted diets compared to low fat diets. There are three possible explanations. First, there might be greater energetic costs associated with metabolic interconversions of nutrients on carbohydrate restricted diets. Second, individuals on a lower carbohydrate diet may have higher energy expenditure due to a greater resting metabolic rate and/or greater levels of physical activity. A final possibility is that lower weight loss is due to the selective under-reporting of dietary intake in individuals randomized to low fat diets. This latter explanation is not likely as this finding has been observed in numerous randomized controlled trials.

   Diet induced thermogenesis may have a small contribution to the metabolic advantage of carbohydrate restricted diets. It accounts for 5-15% of total energy expenditure. The energetic costs to metabolize macronutrients vary from 2.5% with dietary fat, 7-15% with carbohydrate and 28-35% with protein. One study found that energy expenditure was 4% higher in a diet containing 30% compared to 10% of calories from protein. Thus the modest increase in energy expenditure due to a higher protein intake would not likely be enough to account for the metabolic advantage of carbohydrate restricted diets.

   Physical activity is the greatest modifiable source of energy expenditure. The hypothesis that the metabolic advantage of carbohydrate restricted diets could explain lower insulin levels associated with spontaneous increases in physical activity has received scant attention. This hypothesis is based on a number of well established observations. First, type II diabetics taking exogenous insulin have decreases in energy expenditure and weight gain. When insulin levels are lowered through carbohydrate restriction or pharmacotherapy there is an attendant loss of fat mass and some evidence for a modest increase in energy expenditure. A short study of obese individuals found that a ketogenic, low carbohydrate diet with a 30% decrease in insulin resistance was associated with a 20% increase in resting energy-expenditure, though physical activity was not assessed in this study. Similarly, in a 6 month randomized trial of obese women, those on the carbohydrate restricted diet had a non-significant 5% increase in resting energy expenditure per kg of body weight compared to baseline. This study also assessed physical activity using pedometers and found no difference in steps/day between the carbohydrate restricted group and the low-fat group despite a 3.7kg greater weight loss in the former and no difference in reported caloric intake between groups. Measurement of physical activity in free-living individuals is complex. Pedometers are an objective assessment of physical activity but are unable to assess intensity, frequency and duration of activity. They are also unsuitable for estimation of energy expenditure.

   In summary, intensive lifestyle interventions reduce the incidence of type II diabetes in individuals with metabolic syndrome. Central to the therapeutic effect of these interventions is weight loss. There is a lack of consensus over what constitutes 'best practices' for lifestyle interventions. Physical activity is associated with numerous health benefits but is not an efficacious prescription for weight loss or weight maintenance. Moreover, the optimal dietary prescription is controversial; some experts suggest individuals with MetS should restrict their dietary fat intake while other experts suggest dietary carbohydrate should be restricted. This controversy in dietary prescription is reflected in the positions of major medical organizations. The American Diabetes Association has endorsed carbohydrate restriction for weight loss since 2008. The Canadian Diabetes Association, however, favours lower glycemic index foods and the restriction of dietary fat. Despite the equivocal evidence, a low fat, calorie restricted diet coupled with increased physical activity are considered the standard lifestyle interventions for MetS.
2. OBJECTIVES This protocol has three aims. First, the investigators hypothesize that adherence to a lower carbohydrate diet in individuals with MetS, resulting in lower insulin resistance; will cause an increase in levels of spontaneous physical activity, independent of changes in weight. Second, the investigators will examine changes in cardiometabolic risk factors (ApoB, TG, HDL, blood pressure, CRP) when individuals are randomized to either a carbohydrate restricted diet or a low fat/high carbohydrate diet. Finally, the investigators will interview a sub-sample of participants from both study arms (5 in each arm) to conduct open-ended interviews to better understand quality of life issues with respect to the dietary assignment or lifestyle intervention.
3. RESEARCH PLAN Our group has generated cross-sectional data showing a clinically meaningful association between higher carbohydrate intake and lower physical activity, assessed by accelerometer in glucose intolerant individuals. The limitation of these findings relate to the inability to assess causality; that is, if carbohydrate restriction causes increases in physical activity. The strength of the ACTout study is its ability to delineate causal direction using a prospective design and randomization to control for known and unknown confounders.

Study design and participants: Study participants will be randomized to an ad lib carbohydrate restricted group or a low fat, calorie reduced diet for 6 months. The investigators will recruit individuals with metabolic syndrome (MetS) from St. Paul's Metabolic Syndrome Program. Inclusion criteria include a diagnosis of MetS defined as an increased waist circumference and two or more of the following: fasting blood sugar greater than 5.6 mmol/L, fasting triglycerides greater than 1.7 mmol/L, high density lipoprotein (HDL) less than 1.0 mmol/L in men and less than 1.3 mmol/L in women and blood pressure greater than 135/85 or on antihypertensive medication. Potential participants will be excluded if they are following a weight reducing diet, are abusing alcohol or other psychoactive substances, are on psychiatric medication associated with weight gain or have plans to travel during the study period.

Sample size calculation: To calculate sample size the investigators used cross-sectional data with accelerometer measured physical activity and excellent quantitative measures of diet. The investigators assumed a 15% difference in calories consumed as carbohydrates between the dietary treatments. With a significance value of p < 0.05 (two sided test) the investigators found that 27 participants would be required in each group to detect a significant difference in accelerometer measured intensity of activity. To account for possible attrition the investigators will overestimate the sample size by 10 in each arm. The investigators will recruit 72 individuals with 36 in each arm. Based on our sample size calculation, the investigators expect to detect time and diet based differences in addition to a diet*time interaction.

Recruitment strategy: The investigators will recruit individuals with metabolic syndrome from the Metabolic Syndrome Program. Flyers will be posted in the waiting room and the examination rooms of the Program. Flyers will also be given to the administrative assistants responsible for intake of participants into the Program who may choose to notify participants of the study. If a potential participant expresses interest the coordinator will explain the study in sufficient detail to enable informed consent. To assess diet prior to inclusion into the study the investigators will ask potential participants to complete a 3 day diet history and wear the accelerometer for 7 days to ensure that they are not already following a weight reducing diet and to assess baseline physical activity. Individuals compliant with both the dietary recall and baseline assessment of physical activity will be randomized into one of the two dietary assignments.

Randomization: The investigators will use block randomization to prevent the biasing of the randomization process. After each block of subjects is enrolled, the investigators will use a computerized randomization program to randomly assign participants to one of the two dietary assignments. Due to the difficulty in concealing the dietary assignment, the randomized trial will not be blinded; as both researchers and participants will be aware of their dietary assignment. To minimize the contamination of study groups, individual and group sessions will be scheduled at different times.

Carbohydrate restricted diet: Participants will be instructed to restrict carbohydrate consumption to < 20 grams/day while not restricting their caloric intake. Participants will be encouraged to consume vegetables with low carbohydrate content every day including 2 cups of salad greens and 1 cup of vegetables 'that grow above the ground'. One of the physiologic changes associated with a low carbohydrate intake is a loss of salt through the urine. If salt is not replaced participants may experience headaches, nausea, dizziness, lethargy and constipation. Participants will be counselled to increase their salt intake. This has been shown to correct the natiuresis associated with carbohydrate restriction which can cause the aforementioned side effects. Participants will be advised to continue their baseline level of physical activity.

Control group: The control group will be randomized to the intensive lifestyle intervention currently used by the Healthy Heart Program at St. Paul's Hospital to reduce symptoms associated with metabolic syndrome. Participants will be instructed to replace high fat, energy dense foods with foods rich in whole grains, fruits and vegetables. The macronutrient distribution of this diet will be approximately 55% carbohydrate, 15% protein and 30% fat. Individuals will also be instructed to reduce sodium intake to <2300 mg/day and in individuals with hypertension, <1500 mg/day. At the end of the study, participants will have the option to continue on either of the study diets.

Methods to ensure compliance to the dietary assignment: The study coordinator will facilitate activities to support compliance to the dietary assignment, either one-on-one or in a group setting. Group meetings will reinforce compliance by sharing cooking tips, behaviour modification and relapse prevention strategies. In the one-on-one sessions, the study coordinator will review 3 day food records and discuss strategies to increase compliance. Participants from both groups will meet with their clinician after 3 months to assess health indicators and to assure participants of the safety of their dietary assignment.

Qualitative interviews: The investigators will conduct hour long open-ended interviews with 8-10 participants from the study to understand the lived experience of a prudent diet and a carbohydrate restricted diet. Interviews will be recorded and transcribed. The investigators will use grounded theory to look for theories which emerge from the data as opposed to having interpreting the data with an a priori analysis. The investigators will then assign descriptive categories to themes which emerge from the data, such themes could include: effect of their diet on diabetes, perceptions of hunger, mood etc. These descriptive categories will then be placed into thematic categories and analyzed in light of the existing of the literature.

Measurement of body composition and estimation of resting energy expenditure:

The investigators will use bioelectrical impedance to assess body composition at baseline and at 6 months. Bioelectrical impedance has been shown to provide a reasonable assessment of body composition compared to DXA, which is considered a gold standard. The investigators will normalize fat mass and fat-free mass to height by using a fat-mass index and a fat-free mass index (kg/m2), respectively. Height will be measured with a stadiometer at baseline. Waist circumference will be assessed at baseline and at 6 months, after exhalation, using a flexible tape measure half way between the hip bone and the lowest rib. The investigators will estimate energy expenditure using previously published equations which take into account fat-free mass, fat mass, gender and age.

Questionnaire: The investigators will use the Applied Health Indicators Questionnaire and the Patient Health Questionnaire, to collect relevant health information from the patient. These self-administered questionnaires will be completed at baseline, 3 and 6 months.

Physical activity assessment: Participants will wear an accelerometer to assess physical activity at baseline and week of every month for 6 months. An accelerometer is a small electronic monitor worn on the waist that measures vertical accelerations and is thus considered an objective measure of physical activity. Patients will be instructed to wear the accelerometer during waking hours for 1 week of every month, exclusive of time spent bathing or when in water. Data will be downloaded in one-minute epochs and categorized as light, moderate or vigorous activity. Days will be excluded when the accelerometer is worn for less than 80% of the average time worn on the other days. The investigators will estimate activity-based energy expenditure using previously validated equations. As accelerometers do not capture activity associated with cycling, swimming or skiing the investigators will ask participants about the number of times they did these activities in the period that they wore the accelerometer.

Cardiometabolic indices: Blood samples will be drawn and placed in individually labelled tubes with EDTA, centrifuged immediately and stored at -70°C. As changes in insulin action are central to our hypothesis the investigators will assess two distinct aspects of insulin metabolism in this study, insulin secretion and insulin resistance. The investigators will assess insulin resistance using HOMA assessment of insulin resistance calculated from fasting insulin and fasting glucose. The investigators will assess the concentration of C-peptide, a cleavage product related to insulin synthesis that is synthesized in equimolar concentrations to insulin. As C-peptide has a longer half-life than insulin, it can be used a marker of insulin secretion from the pancreas. Blood Pressure will be assessed at baseline, 3 and 6 months using BP-TRU monitors. Lipid, lipoprotein and C-reactive protein levels will be measured at baseline, 3 and 6 months. Total cholesterol, triglyceride, high-density lipoprotein cholesterol and apolipoprotein B will be measured using previously described methods. LDL-chol levels will be calculated using the Friedewald formula for patients whose plasma triglyceride level is less than 4 mmol/L. β-hydroxybutyrate will also be assessed in both groups at the aforementioned time points and will be used as a biomarker of adherence to a carbohydrate restricted diet. The investigators will also assess serum Leptin and uric acid at baseline and 6 months.

Statistical analyses: The investigators will use two different approaches to analyze the data. First the investigators will use an intention to treat analysis using baseline values to impute missing data in participants who may drop-out of the study. The investigators will also examine the effect of the dietary assignment on outcomes in participants who were compliant with their dietary assignment. Baseline characteristics will be compared between the two groups using t tests. The investigators will examine three inter-related dependent variables, capturing different aspects of physical activity, in the analysis strategy. First, the investigators will examine the association between dietary assignment and changes in accelerometer variables. The investigators will also examine time spent in moderate-to-vigorous physical activity and activity based energy expenditure. As activity based energy will be estimated from accelerometer , the investigators will not consider it a unique comparison. The investigators will thus set the level of statistical significance at p<0.025 to adjust for multiple comparisons. The investigators will obtain differences in key variables such as physical activity and change in insulin concentration. To assess the effects of the dietary assignment on physical activity, the investigators will use three-way repeated-measures ANOVA, including change in body weight in the model with time as the repeated factor.

ELIGIBILITY:
Inclusion Criteria:

* presence of metabolic syndrome by International Diabetes Foundation criteria
* referral to metabolic syndrome program at St. Paul's Hospital
* age > 19 years

Exclusion Criteria:

* unwillingness to participate in research study
* unwillingness to comply with dietary intervention
* following a weight reducing diet
* abusing alcohol or other psychoactive substances
* on psychiatric medication associated with weight gain
* plans to travel during the study period
* food allergies or intolerances that will interfere with their adherence to either of the study diets

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
changes in physical activity from baseline | 3 and 6 months
  1. activity counts per minute;
  2. time spent in light and moderate to vigorous physical activity;
  3. activity based energy expenditure using previously validated equations

SECONDARY OUTCOMES:
Change in lipids from baseline | 3 and 6 months
  total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, apolipoprotein B, apolipoprotein A1
change in renal function from baseline | 3 and 6 months
  creatinine, urine microalbumin/creatinine ratio, serum and urine NGAL

CONTACTS AND LOCATIONS:
Overall Officials: Sammy Chan, MD, Principal Investigator — St. Paul's Hospital, Vancouver
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada